CLINICAL TRIAL: NCT00849771
Title: Multicenter Prospective Study of Operative and Non-operative Treatment for Scapula Fractures
Brief Title: Operative Versus Nonoperative Treatment for Scapula Fractures
Status: Withdrawn | Type: Observational
Why Stopped: Joined another larger group of same study
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, William Obremskey, Chief of Orthopedic Trauma, Vanderbilt University
Other Study IDs: 080160
Record Dates: First submitted 2009-02-20; First posted 2009-02-24 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Scapula Fracture; Clavicle Fracture
Keywords: Displaced Scapula Fracture; Scapula Fracture; Extraarticular Scapula Fractures; Clavicle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Operative Treatment (Open Reduction Internal Fixation)
- 2: Non-operative/Conservative Care

SUMMARY:
The purpose of this study is to contrast and evaluate the functional outcome of patients with operative vs. nonoperative treatment of scapula fractures. The specific aim of this project is to monitor the return to function of patients in both the operative and nonoperative cohorts.

The potential impact is a clearer set of choices in treatment options for this type of injury.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years of Age or Older
* Displacement of glenoid neck and scapula body of greater than 2 cm
* Angular deformity between the fracture fragments of greater than 45 degrees.
* A combination of displacement greater than 1.5 cm AND angulation greater than 30 degrees
* A glenopolar angle less than 22 degrees
* A Double Lesion of the Superior Shoulder Suspensory Complex (SSSC)

Exclusion Criteria:

* Age Less Than 18 years Old
* Brachial Plexus Injury
* Traumatic Brain Injury or Cognitive Disability preventing participation in the consent or post injury rehabilitation
* Spinal cord injuries resulting in paraplegic, quadriplegic disabilities or permanent ipsilateral peripheral nerve damage
* Ipsilateral Upper Extremity Injury
* Previous Shoulder Surgery
* Insufficient English proficiency to complete the DASH Questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject population will include patients seen at participating facilities for the care of scapula fractures, who are 18 years of age or older, meet inclusion/exclusion criteria and are willing to consent.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-03; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William T. Obremskey, MD, MPH, Principal Investigator — Vanderbilt University Medical Center; Peter Cole, MD, Principal Investigator — University of Minnesota
Locations (1):
- Vanderbilt Orthopaedic Institute, Vanderbilt University Medical Center, Nashville, Tennessee, United States